



## **Research Title:**

Periotome Versus Peizotome as an Aid of Atraumatic Extraction.

**Consent Form** 

**Date:** 

Septemper 1, 2019





## **Participation Consent Form**

| l | signed below |
|---|---|
| Authorize the doctor to perform the extraction of tooth number ( or Piezome as a new techniques of atraumatic simple extraction and the reduction of procedure and after the procedure pain. A been explained to me and I accept my participation in this study | for the preservation of bone<br>all possible complications have |
| Signature: | |
| Date: | |